CLINICAL TRIAL: NCT01671124
Title: Phase IIa Study of Antidepression Use Natural Plants Extracted of Soline Capsule.
Brief Title: The Study of Antidepressant Properties and Safety of Fer-01(Soline®) on the Patients With Depression
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Medical University Hospital (Other)
Collaborators: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Fer-01
Record Dates: First submitted 2012-08-15; First posted 2012-08-23 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-08

CONDITIONS: Major Depressive Disorder
Keywords: TG; TC; HDL; LDL; Albumin; Hemoglobin; Hematocrit; Uric acid; Sodium; Potassium; Calcium
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Fluoxetine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Soline capsule: Salvia divinorum, Lycium, Chenpi and Dihuang
  Interventions: Other: Soline capsule

INTERVENTIONS:
Other: Soline capsule
  Other Names: prozac

SUMMARY:
Considering the potential modulatory effects of Salvia divinorum, Lycium, Chenpi and Dihuang supplementation on mood, this study is a clinical study of Soline® (product mixed with Salvia divinorum, Lycium, Chenpi and Dihuang ) supplementation to investigate the effect of attenuating the occurrence of depression. The study will enroll 100 patients who meet the inclusion and exclusion criteria. The trial will be concluded when a total of evaluable 80 patients (40 patients in each treatment group).

DETAILED DESCRIPTION:
Depression is one of the major metal disorders associated with symptoms such as regular negative moods, decreased physical activities, feeling of helplessness, and cognitive deficits. According to the seminal "burden of disease" study by World Health Organization (WHO) has predicted that by 2030 depression will be the second leading cause of disease. The Diagnostic and Statistical Manual of Mental Disorders (DSM) is the American Psychiatric Association's standard reference for psychiatry which includes over 400 different definitions of mental disorders. Selective and reversible monoamine oxidase inhibitor, selective serotonin reuptake inhibitors or serotonin and noradrenaline reuptake inhibitors are the typical antidepressants usually. Unfortunately, current drug therapies for depression are not ideal. Most of the drugs are synthetic nitrogen-bearing compounds which have inevitably some serious adverse-effects such as causing cardiovascular disease, insomnia and ovarian teratomas. Hence, there is an urgent need for the research and development of more effective antidepressants without any/ with minor adverse-effect. Up to the present, many Chinese medicinal plants have been successfully used to treat sentimental diseases, which is similar to depression in the Western medicine. Shamans of the Mazatec people of Oaxaca, Mexico have used Salvia divinorum for at least centuries in ethnomedical practices including spiritual healing and divinorum. Salvia divinorum contains the known psychoactive constituent salvinorin A, which is a trans-neoclerodancediterpenoid and a к-opioid agonist with no activity at the 5-HT2A serotonin receptor, making it an ideal agent for antidepressant. Salvia divinorum use occurring in Europe and Japan, and survey research suggests that user claim positive after-effects. Lycium, Chenpi ( Citrus reticulate Blanco ) and Dihuang ( Rehmannia glutinosa ) were widely used in the vast majority of Chinese medicine prescription to treat mental disease, for example, Lily Bulb Decoction to Preserve the Lung ( Lycium and Dihuang ) from Analytic Collection of Medical Formula , Spirit-quieting Decoction ( Chenpi ) form Restoring Health from Tens of Thousands of Diseases. Considering the potential modulatory effects of Salvia divinorum, Lycium, Chenpi and Dihuang supplementation on mood, this study is a clinical study of Soline® (product mixed with Salvia divinorum, Lycium, Chenpi and Dihuang ) supplementation to investigate the effect of attenuating the occurrence of depression.

ELIGIBILITY:
Inclusion Criteria:

•Clinical diagnosis of major depressive disorder

Exclusion Criteria:

* Pregnancy and nursing
* Schizophrenia spectrum disorder
* Manic depressive disorder
* Bipolar disorder
* Anxiety Disorder
* Abnormal biochemistry analysis value:( AST and ALT≧triple the upper limit of normal)；
* Serum creatinine>2mg/dl
* BUN>40mg/dL
* Total bilirubin>2.0mg/dL
* Hematocrit<30
* White blood count≧15000
* High sensitivity to this product
* The diseases will influence of results: pulmonary tuberculosis, uncontrolled diabetes, uncontrolled hypertension, serious infection and critical cardiovascular, liver, kidney disease.
* Alcohol abuse or drug abuse
* Attended the other study in last 4 weeks
* Attempted suicide or self-injurious

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: community sample, residents of Taiwan
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-07 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
DSM-IV | Day 1 and up to 6 weeks
  diagnosis of major depressive disorder according to DSM-Ⅳ has change

SECONDARY OUTCOMES:
analysis of inflammation cytokine | Day 1 and up to 6 weeks
  Laboratory examination parameters ( TNF-a,IL-6, TGF-b1)
analysis of basic biochemical | Day 1 and up to 6 weeks
  The incidence of hepatic and renal adverse events(GOT, GTP, BUN, creatinine...)
Fatty acid composition | Day 1 and up to 6 weeks
  Fatty acid composition is measure with gas chromatography.

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Yi Huang, Ph.D, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Mecical University Hospital, Taipei, Taiwan, Taiwan